CLINICAL TRIAL: NCT03486522
Title: Screening for Sexually Transmitted Diseases (STDs) in Women Admitted in Family Planning, Lariboisière Hospital, for a Termination of Pregnancy: a Prospective Systematic Survey.
Brief Title: STD Screening in Women Admitted in Family Planning for a Termination of Pregnancy
Acronym: DEP-IST-IVG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hopital Lariboisière (Other)
Responsible Party: Principal Investigator, Célia Lloret-Linares, MD PhD, PI, Hopital Lariboisière
Other Study IDs: 2018-A00144-51
Record Dates: First submitted 2018-03-18; First posted 2018-04-03 (Actual); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: STD
Keywords: termination of pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Epidemiology of Sexually Transmitted Diseases (STDs) in women admitted in a Family Planning for a termination of pregnancy is poorly defined currently in France. Only one bi-centre study (Bourgeois-Nicolaos, 2015), performed in two Family Planning suburban centres located within University Hospital (Assistance Publique-Hôpitaux de Paris), found high prevalence: C. trachomatis 15.1%, N. gonorrhoeae 3.1%. Moreover, heterogeneity can occur between centres. In students in Sweden, 26% had one or several previous STDs, mainly C. trachomatis and Human Papilloma Virus (HPV). Having previously a termination of pregnancy was a risk factor of STDs. Systematic screening for STDs in Women Admitted in Family Planning for a Termination of Pregnancy appears thus a logical strategy.

DETAILED DESCRIPTION:
Epidemiology of Sexually Transmitted Diseases (STDs) in women admitted in a Family Planning for a termination of pregnancy is poorly defined currently in France. Only one bi-centre study (Bourgeois-Nicolaos, 2015), performed in two Family Planning suburban centres located within University Hospital (Assistance Publique-Hôpitaux de Paris), found high prevalence: C. trachomatis 15.1%, N. gonorrhoeae 3.1%. Moreover, heterogeneity can occur between centres. In students in Sweden, 26% had one or several previous STDs, mainly C. trachomatis and Human Papilloma Virus (HPV). Risk factors in univariate analysis were tobacco smoking, a previous termination of pregnancy, lack of vaccination against HPV, having sexual intercourse precociously, number of sexual partners, anal sex, having sexual intercourse without consent, having unprotected sex during last intercourse. Risk factors in multivariate analysis were a previous termination of pregnancy, lack of vaccination against HPV, number of sexual partners, having sexual intercourse without consent, having unprotected sex during last intercourse. Systematic screening for STDs in Women Admitted in Family Planning for a Termination of Pregnancy appears thus a logical strategy.

In a previous study performed in Emergency Dpt in an University Hospital (Assistance Publique-Hôpitaux de Paris), screening patients born in sub-Saharan Africa, French Indies and French Guyana, prevalence 1.8% (6 times national prevalence), 7.8% and 3.6% for HIV, HBV and HCV was found respectively. Ile-de-France is the area of France with the highest HBV prevalence (133/100 000); moreover, most women with HBsAg positive are of child-bearing age. From the 24,000 women with HBsAg positive 18-39 years old, only 5700 (24%) are aware of their status. Similarly, Ile-de-France is the area of France with the highest HCV prevalence (109/100 000), with women 20-29 and 30-39 years old accounting for 15% each. HCV nationale prévalence is 3.1% in people born in sub-Saharan Africa, 1.4% in people born in Asia, 10.2% in people born in Middle-East.

ELIGIBILITY:
Inclusion Criteria: Women of age or not coming for a termination of pregnancy able to give a written consent for the survey

Exclusion Criteria:Women coming for another reason than a termination of pregnancy

* Not able to to give a written consent for the Survey
* Women with legal guardian
* Women who refused to take part to the survey

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All women, of age or not, with a pregnancy less than 14 weeks of amenorrhae, who came to the family planning centre of Obstetrics Dpt, Lariboisière Hospital, for a termination of pregnancy, able to give a written consent for the Survey.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-03-16 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
STDs prevalence | Up to 30 days after termination of pregnancy (period of follow-up)
  Prevalence of STDs (C trachomatis, N gonorrhoae, T pallidum, HIV, HBV, HCV, HPV) in women in a family planning centre

CONTACTS AND LOCATIONS:
Overall Officials: Pierre O Sellier, M.D., Ph.D., Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Family Planning Centre, Obstetrics Dpt, Lariboisière Hosp,, Paris, Île-de-France Region, France